CLINICAL TRIAL: NCT01070212
Title: Effects of Gum Chewing on Appetite and Digestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Prof. Foods and Nutrition, Purdue University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: R01DK079913-2; R01DK079913 (NIH); 0911008653 (Other: Purdue University)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: The Null Hypothesis is That Food Rheology Will Have no Effect on These Indices; The Alternate Hypothesis is That Increased Mechanical Stimulation Will Result in Stronger Satiation/Satiety and Reduced Energy Intake; It is Hypothesized That the Effects of Mastication Will be Less Evident in Obese Compared to Lean Individuals
Keywords: human, chewing, appetite,

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- soft gum (Experimental): . Participants will either chew nothing or chew one of the two gum varieties (flavorless soft or hard) at a constant rate (determined by a metronome) for 15 minutes while sipping apple juice through a straw. Appetite will be measured continuously via a slide potentiometer attached to a 100mm gLMS scale. The juice will provide 10% of the participants estimated daily energy requirement (i.e., equal to 1-2 servings of most commercial snacks). It will also contain 10g of lactulose (a soluble, non-absorbable carbohydrate used to assess gastric transit time via analyses of breath hydrogen) and acetaminophen (a marker for gastric emptying).
  Interventions: Other: soft gum
- firm gum (Experimental): . Participants will either chew nothing or chew one of the two gum varieties (flavorless soft or hard) at a constant rate (determined by a metronome) for 15 minutes while sipping apple juice through a straw. Appetite will be measured continuously via a slide potentiometer attached to a 100mm gLMS scale. The juice will provide 10% of the participants estimated daily energy requirement (i.e., equal to 1-2 servings of most commercial snacks). It will also contain 10g of lactulose (a soluble, non-absorbable carbohydrate used to assess gastric transit time via analyses of breath hydrogen) and acetaminophen (a marker for gastric emptying).
  Interventions: Other: firm gum
- no gum (Experimental): . Participants will either chew nothing or chew one of the two gum varieties (flavorless soft or hard) at a constant rate (determined by a metronome) for 15 minutes while sipping apple juice through a straw. Appetite will be measured continuously via a slide potentiometer attached to a 100mm gLMS scale. The juice will provide 10% of the participants estimated daily energy requirement (i.e., equal to 1-2 servings of most commercial snacks). It will also contain 10g of lactulose (a soluble, non-absorbable carbohydrate used to assess gastric transit time via analyses of breath hydrogen) and acetaminophen (a marker for gastric emptying).
  Interventions: Other: no gum

INTERVENTIONS:
Other: soft gum — . Participants will either chew nothing or chew one of the two gum varieties (flavorless soft or hard) at a constant rate (determined by a metronome) for 15 minutes while sipping apple juice through a straw. Appetite will be measured continuously via a slide potentiometer attached to a 100mm gLMS scale. The juice will provide 10% of the participants estimated daily energy requirement (i.e., equal to 1-2 servings of most commercial snacks). It will also contain 10g of lactulose (a soluble, non-absorbable carbohydrate used to assess gastric transit time via analyses of breath hydrogen) and acetaminophen (a marker for gastric emptying).
  Arms: soft gum
Other: firm gum — . Participants will either chew nothing or chew one of the two gum varieties (flavorless soft or hard) at a constant rate (determined by a metronome) for 15 minutes while sipping apple juice through a straw. Appetite will be measured continuously via a slide potentiometer attached to a 100mm gLMS scale. The juice will provide 10% of the participants estimated daily energy requirement (i.e., equal to 1-2 servings of most commercial snacks). It will also contain 10g of lactulose (a soluble, non-absorbable carbohydrate used to assess gastric transit time via analyses of breath hydrogen) and acetaminophen (a marker for gastric emptying).
  Arms: firm gum
Other: no gum — . Participants will either chew nothing or chew one of the two gum varieties (flavorless soft or hard) at a constant rate (determined by a metronome) for 15 minutes while sipping apple juice through a straw. Appetite will be measured continuously via a slide potentiometer attached to a 100mm gLMS scale. The juice will provide 10% of the participants estimated daily energy requirement (i.e., equal to 1-2 servings of most commercial snacks). It will also contain 10g of lactulose (a soluble, non-absorbable carbohydrate used to assess gastric transit time via analyses of breath hydrogen) and acetaminophen (a marker for gastric emptying).
  Arms: no gum

SUMMARY:
One obvious property difference between energy-yielding beverages and solid foods is the oral mechanical processing required to prepare the two food forms for swallowing. Considerable human data are consistent with a contribution of mechanical stimulation to appetite suppression. However, no study has isolated this property and assessed its influence on ingestive behavior in humans. This is the aim of the present study. The null hypothesis is that food rheology will have no effect on these indices. The alternate hypothesis is that increased mechanical stimulation will result in stronger satiation/satiety and reduced energy intake. Further, it is hypothesized that the effects of mastication will be less evident in obese compared to lean individuals.

ELIGIBILITY:
Inclusion Criteria:

* body mass index 18 -25 or 30-35 kg/ m2 good health not initiating or terminating the use of medications reported to affect appetite or body weight during the proposed study period stable activity level (no deviation > 1X/wk @ 30 min/session) no eating disorder (score <20 of the Eating Attitude Test (EAT-26) no allergies to test foods. not glucose intolerant or diabetic (based on fasting blood glucose between 70-99mg/dl (3.9-5.5mmol/l as recommended by the American Diabetes Association.) no history of GI pathology and self-reported consumer of breakfast and lunch.

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Effects of mastication on appetite. | 12 hours
  Effects of varying chewing intensity on self-rated hunger, fullness, desire to eat and thirst.

SECONDARY OUTCOMES:
Endocrine response | 4 hours
  Effects of varying chewing intensity on serum/plasma GLP-1, Ghrelin, CCK, Insulin.
Blood chemistries | 4 Hours
  Effects of varying chewing intensity on lipid profiles and glucose.

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States